CLINICAL TRIAL: NCT00963469
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Investigating the Clinical Effect of Montelukast in Patients With Seasonal Allergic Rhinitis Over a 4-Week Treatment Period-Fall 2001
Brief Title: Montelukast in Seasonal Allergic Rhinitis: Fall 2001 Study (0476-240)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-240; MK0476-240; 2009_647
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast sodium
- 2 (Active Comparator): loratadine
  Interventions: Drug: Comparator: loratadine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: montelukast sodium — montelukast 10 mg tablet orally once daily in the morning for 4 weeks
  Arms: 1
Drug: Comparator: loratadine — loratadine 10 mg tablet orally once daily in the morning for 4 weeks
  Arms: 2
Drug: Comparator: placebo — placebo tablet orally once daily in the morning for 4 weeks
  Arms: 3

SUMMARY:
This is a study to evaluate the treatment effect of montelukast 10 mg taken in the morning, versus placebo, in patients with seasonal allergic rhinitis. Loratadine is included in the study as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of seasonal allergic rhinitis that worsens during the study season
* Patient is a nonsmoker
* Patient is in good health physical and mental health

Exclusion Criteria:

* Patient is hospitalized
* Patient is a woman who is < 8 weeks postpartum or is breastfeeding
* Patient plans to move or vacation away during the study
* Patient has had any major surgery with in past 4 weeks
* Patient is a current or past abuser of alcohol or illicit drugs

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1079 (Actual)
Dates: Start 2001-08; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] van Adelsberg J, Philip G, Pedinoff AJ, Meltzer EO, Ratner PH, Menten J, Reiss TF; Montelukast Fall Rhinitis Study Group. Montelukast improves symptoms of seasonal allergic rhinitis over a 4-week treatment period. Allergy. 2003 Dec;58(12):1268-76. doi: 10.1046/j.1398-9995.2003.00261.x. PMID 14616102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-seven study centers in the United States.
  Prime Therapy Period: August 2001 to November 2001
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined daytime nasal symptoms score during the run-in period were excluded from randomization.
Groups:
- Placebo: Montelukast matching-image placebo tablet and Loratadine matching-image placebo tablet orally once daily in the morning for 4 weeks
- Montelukast: Montelukast 10-mg tablet and Loratadine matching-image placebo tablet orally once daily in the morning for 4 weeks
- Loratadine: Montelukast matching-image placebo tablet and Loratadine 10-mg tablet orally once daily in the morning for 4 weeks
Period: Overall Study
Arm/Group | Placebo | Montelukast | Loratadine
Started | 451 | 448 | 180
Completed | 410 | 420 | 170
Not Completed | 41 | 28 | 10
Not completed — Adverse Event | 15 | 11 | 1
Not completed — Lack of Efficacy | 10 | 7 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Protocol Violation | 5 | 5 | 3
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Pre-randomization Adverse Event | 1 | 2 | 0
Not completed — Moved | 1 | 0 | 0
Not completed — Site closed (local pollen Season ended) | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast | Loratadine | Total
Number analyzed (Participants) | 451 | 448 | 180 | 1079
Age, Continuous [Mean (Full Range); unit: years] | 35.9 [15 to 82] | 35.5 [15 to 82] | 38.7 [15 to 79] | 36.2 [15 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 301 | 119 | 721
  Male | 150 | 147 | 61 | 358
Composite Symptoms Score [Mean (Standard Deviation); unit: Scores on a scale] — Composite Symptoms Scores were computed as the average of Daytime Nasal Scores (Score 0 (best) to 3 (worst)) and Nighttime Symptoms Scores [Score 0 (best) to 3 (worst)].
  Scores on a scale | 1.94 (0.46) | 1.98 (0.47) | 2.03 (0.46) | 1.97 (0.46)
Daytime Eye Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Daytime Eye Symptoms scores. Patients were asked to rate each of the 4 eye symptoms of tearing, itchy, red, and puffy eyes daily on a 4-point scale [Score 0 (best) to 3 (worst)]. The average of the 4 individual eye symptoms scores was reported as the Daytime Eye Symptoms Score.
  Scores on a scale | 1.61 (0.81) | 1.64 (0.73) | 1.64 (0.78) | 1.63 (0.77)
Daytime Nasal Symptoms Score [Mean (Standard Deviation); unit: Scores on a scale] — Daytime Nasal Symptoms Score. Patients were asked to rate each nasal symptom of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4-point scale [Score 0 (best) to 3 (worse)]. The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal Symptoms Score.
  Scores on a scale | 2.16 (0.44) | 2.20 (0.46) | 2.23 (0.44) | 2.19 (0.45)
Nighttime Symptoms Score [Mean (Standard Deviation); unit: Scores on a scale] — Nighttime Symptoms Score. Patients were asked to rate each symptom of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings daily on a 4-point scale [Score 0 (best) to 3 (worse)], and the average score of the 3 symptoms was reported as the Nighttime Symptoms Score.
  Scores on a scale | 1.65 (0.64) | 1.69 (0.64) | 1.77 (0.63) | 1.69 (0.64)
Rhinoconjunctivitis Quality of Life Score [Mean (Standard Deviation); unit: Scores on a scale] — Patients completed a Rhinoconjunctivitis Quality-of-Life Questionnaire-28 questions on a 7-point scale [0(best) to 6(worst)] across 7 domains: activity,sleep,non-nose/eye symptoms,practical problems,nasal symptoms, eye symptoms, and emotions. The scores for each domain were averaged, then scores for the 7 domains were averaged for an overall score.
  Scores on a scale | 3.37 (1.02) | 3.41 (1.00) | 3.46 (1.08) | 3.40 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score Over First 2 Weeks of Treatment Period
Description: Mean change from baseline in Daytime Nasal Symptoms Score.
  Patients were asked to rate each nasal symptom of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4- point scale [Score 0 (best) to 3 (worse)]. The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal Symptoms Score.
Time Frame: Baseline and first 2 Weeks of treatment period (from randomization through the end of Week 2)
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement through the first 2 weeks of treatment were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 448 | 445 | 180
Scores on a scale | -0.23 [-0.28 to -0.18] | -0.33 [-0.37 to -0.28] | -0.45 [-0.52 to -0.37]

2. Secondary Outcome: Mean Change From Baseline in Nighttime Symptoms Score Over First 2 Weeks of Treatment Period
Description: Mean change from baseline in Nighttime Symptoms Score.
  Patients were asked to rate each symptom daily on a 4-point scale [Score 0 (best) to 3 (worse)], and the combined score of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings was reported as the Nighttime Symptoms Score.
Time Frame: Baseline and first 2 Weeks of treatment period (from randomization through the end of Week 2)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 448 | 445 | 180
Scores on a scale | -0.18 [-0.23 to -0.14] | -0.28 [-0.32 to -0.23] | -0.25 [-0.32 to -0.19]

3. Secondary Outcome: Mean Change From Baseline in Composite Symptoms Score (Daytime Nasal and Nighttime Symptoms) Over First 2 Weeks of Treatment Period
Description: Composite Symptoms Scores were computed as the average of Daytime Nasal Scores [Score 0 (best) to 3 (worst)] and Nighttime Symptoms Scores [Score 0 (best) to 3 (worst)].
Time Frame: Baseline and first 2 Weeks of treatment period (from randomization through the end of Week 2)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 448 | 445 | 180
Scores on a scale | -0.21 [-0.25 to -0.16] | -0.30 [-0.35 to -0.26] | -0.36 [-0.43 to -0.30]

4. Secondary Outcome: Mean Change From Baseline in Daytime Eye Symptoms Score Over First 2 Weeks of Treatment Period
Description: Mean change from baseline in Daytime Eye Symptoms scores.
  Patients were asked to rate each of the 4 eye symptom of tearing, itchy, red, and puffy eyes daily on a 4-point scale [Score 0 (best) to 3 (worst)]. The average of the 4 individual eye symptoms scores was reported as the Daytime Eye Symptoms Score.
Time Frame: Baseline and first 2 Weeks of treatment period (from randomization through the end of Week 2)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 448 | 445 | 180
Scores on a scale | -0.18 [-0.23 to -0.14] | -0.28 [-0.33 to -0.23] | -0.33 [-0.41 to -0.26]

5. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis After First 2 Weeks of Treatment
Description: An evaluation by the patient, administered after the first 2 weeks of treatment using a 7-point scale [Score 0 (best) to 6 (worst)], of the change in symptoms as compared to the beginning of the study.
Time Frame: After first 2 weeks of treatment
Population: The primary efficacy analyses were based on the intention-to-treat. Since only 1 measurement was obtained during the treatment period, no missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 447 | 444 | 178
Scores on a scale | 2.73 [2.59 to 2.88] | 2.43 [2.29 to 2.57] | 2.30 [2.08 to 2.52]

6. Secondary Outcome: Physician's Global Evaluation of Allergic Rhinitis After First 2 Weeks of Treatment
Description: An evaluation by the physician, administered after the first 2 weeks of treatment using a 7-point scale [Score 0 (best) to 6 (worst)], of the change in symptoms as compared to the beginning of the study.
Time Frame: After first 2 weeks of treatment
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 434 | 424 | 172
Scores on a scale | 2.75 [2.62 to 2.88] | 2.36 [2.23 to 2.50] | 2.38 [2.18 to 2.59]

7. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality-of-Life Score After First 2 Weeks of Treatment Period
Description: Patients completed a Rhinoconjunctivitis Quality-of-Life Questionnaire-28 questions on a 7-point scale [0(best) to 6(worst)] across 7 domains: activity,sleep,non-nose/eye symptoms,practical problems,nasal symptoms, eye symptoms, and emotions. The scores for each domain were averaged, then scores for the 7 domains were averaged for an overall score.
Time Frame: Baseline and first 2 Weeks of treatment period (from randomization through the end of Week 2)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 448 | 444 | 180
Scores on a scale | -0.55 [-0.65 to -0.45] | -0.85 [-0.94 to -0.75] | -0.85 [-1.00 to -0.70]

ADVERSE EVENTS:
Time Frame: During the 4 week, double-blind treatment period, and up to and including 14 days after the last dose of study therapy.
Description: The number of patients listed in the Adverse Event (AE) tables (448 montelukast group, 180 loratadine group and 451 in placebo group) is the number of patients who received study treatment.
  Although a patient may have had two or more clinical AEs the patient is counted only once in a category. The same patient may appear in different categories.
Arm/Group | Placebo | Montelukast | Loratadine
Serious Adverse Events (participants affected / at risk) | 0/451 | 2/448 | 0/180
Other Adverse Events (participants affected / at risk) | 22/451 | 27/448 | 12/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=451) | Montelukast (N=448) | Loratadine (N=180)
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=451) | Montelukast (N=448) | Loratadine (N=180)
Headache (Nervous system disorders) | 22 | 27 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.